CLINICAL TRIAL: NCT04177043
Title: Educate, Test and Treat Model Towards Elimination of Hepatitis C Infection in Egypt: Feasibility and Effectiveness in 73 Villages
Brief Title: Model Towards Elimination of Hepatitis C Infection in Egypt: Feasibility and Effectiveness in 73 Villages
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: village2015
Record Dates: First submitted 2019-02-20; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (Other)
  Interventions: Diagnostic Test: HCV antibody and hepatitis B surface antigen (HBsAg) rapid diagnostic tests; Drug: DAAs

INTERVENTIONS:
Diagnostic Test: HCV antibody and hepatitis B surface antigen (HBsAg) rapid diagnostic tests — HCV antibody and hepatitis B surface antigen (HBsAg) rapid diagnostic tests
Drug: DAAs — Treatment with different regiments with DAAs

SUMMARY:
Background: The global response to the HCV infection epidemic has been transformed by the availability of low-cost curative short course direct acting antiviral (DAA) therapy. Egypt has one of the highest burdens of HCV infection worldwide, and a large treatment programme, but reaching rural communities represents a major challenge. We report the feasibility and effectiveness of a comprehensive community-based HCV prevention, testing and treatment model in 73 villages across Egypt, with the goal to eliminate infection from all adult villagers.

Methods: An HCV "educate, test and treat" programme was implemented in 73 villages across 7 governorates in Egypt between 06/2015 and 06/2018. The programme model comprised community mobilization facilitated by a network of village promoters to support the education, test and treat campaign as well as fund raising in the local community; a comprehensive testing, linkage to care and treatment of all eligible villagers aged 12 to 80 years using HCV antibody and HBsAg rapid diagnostic tests (RDTs), HCV RNA confirmation of positive cases, staging of liver disease using transient elastography (FibroScan), treatment with 12 or 24 weeks of a direct acting antiviral (DAA) regimen according to national standard of HCV care, and an assessment of cure at 12 weeks after completion of treatment (SVR12); and an education campaign to raise awareness and disseminate messages about safer practices to reduce transmission through public events, promotional materials and house-to-house visits. Key outcomes assessed in each village were: uptake of serological HCV and HBV testing, linkage to assessment and HCV viral load confirmation, uptake of treatment, and SVR12.

DETAILED DESCRIPTION:
Background: The global response to the HCV infection epidemic has been transformed by the availability of low-cost curative short course direct acting antiviral (DAA) therapy. Egypt has one of the highest burdens of HCV infection worldwide, and a large treatment programme, but reaching rural communities represents a major challenge. We report the feasibility and effectiveness of a comprehensive community-based HCV prevention, testing and treatment model in 73 villages across Egypt, with the goal to eliminate infection from all adult villagers.

Methods: An HCV "educate, test and treat" programme was implemented in 73 villages across 7 governorates in Egypt between 06/2015 and 06/2018. The programme model comprised community mobilization facilitated by a network of village promoters to support the education, test and treat campaign as well as fund raising in the local community; a comprehensive testing, linkage to care and treatment of all eligible villagers aged 12 to 80 years using HCV antibody and HBsAg rapid diagnostic tests (RDTs), HCV RNA confirmation of positive cases, staging of liver disease using transient elastography (FibroScan), treatment with 12 or 24 weeks of a direct acting antiviral (DAA) regimen according to national standard of HCV care, and an assessment of cure at 12 weeks after completion of treatment (SVR12); and an education campaign to raise awareness and disseminate messages about safer practices to reduce transmission through public events, promotional materials and house-to-house visits. Key outcomes assessed in each village were: uptake of serological HCV and HBV testing, linkage to assessment and HCV viral load confirmation, uptake of treatment, and SVR12.

ELIGIBILITY:
Inclusion Criteria:

* persons aged between 12 to 80 years across the 73 villages eligible for inclusion in the test and treat program.

Exclusion Criteria:

* aged below 12

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 221855 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
incidince of HCV in population | 3 years
  incidence of HCV hidden population confirmed by Rt-PCR

IPD SHARING:
Plan to Share IPD: No